CLINICAL TRIAL: NCT04687553
Title: Validation of the Chinese Version of the Simplified Evaluation of CONsciousness Disorders (SECONDs)
Brief Title: Validation of the Chinese Version of the SECONDs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hangzhou Normal University (Other)
Responsible Party: Principal Investigator, Jing Wang, Principal Investigator, Hangzhou Normal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2020W356354
Record Dates: First submitted 2020-12-08; First posted 2020-12-29 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Minimally Conscious State; Vegetative State
Keywords: disorders of consciousness; vegetative state; minimally conscious state; consciousness
MeSH Terms: conditions — Persistent Vegetative State; Consciousness Disorders

STUDY DESIGN:
Intervention Model Description: The order of the administration was randomly selected. All patients' total scores assessed by rater A were recorded to test the internal consistency of SECONDs (A1). Meanwhile, to assess the concurrent validity, the scores of the CRS-R were recorded together with SECONDs by rater A on day 1. In order to analyze the test-retest reliability, rater A complete the second evaluation of SECONDs on day 2 (A2).
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with vegetative state (Experimental): Patients with vegetative state were assessed by the SECONDs and CRS-R for two days.
  Interventions: Diagnostic Test: Simplified Evaluation of CONsciousness Disorders (SECONDs)
- Patients with minimally conscious state (Experimental): Patients with minimally conscious state were assessed by the SECONDs and CRS-R for two days.
  Interventions: Diagnostic Test: Simplified Evaluation of CONsciousness Disorders (SECONDs)

INTERVENTIONS:
Diagnostic Test: Simplified Evaluation of CONsciousness Disorders (SECONDs) — All patients were assessed by the Simplified Evaluation of CONsciousness Disorders (SECONDs)

SUMMARY:
The aim of this study was to translate the SECONDs from English into Chinese and determine the validity of this Chinese version

DETAILED DESCRIPTION:
The assessment is of great importance for the management and treatment in patients with disorders of consciousness. The Simplified Evaluation of CONsciousness Disorders is a useful tool to assess consciousness of DOC patients in bedside. The aim of this study was to translate the SECONDs from English into Chinese and determine the validity of this Chinese version. To test internal reliability and inter-rater reliability, both rater A and rater B assess the perception of pain on day 1; and to obtain test-retest reliability, rater A assessed all patients repeatedly on day 2.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 16 years old;
* no administration of neuromuscular blockers or sedation within the 24 hours of enrolment;
* the presence of periods of eye opening (indicating wakefulness and rest cycles);
* a diagnosis of VS or MCS, based on more than 4 times behavioral assessment performed using the Coma Recovery Scale-Revised within 2 weeks.

Exclusion Criteria:

* Coma;
* documented history of prior brain injury;
* psychiatric or neurologic illness;
* neuromuscular blocking agents or sedative drugs administered within the prior 24 hours;
* no documented history of a prior coma, critical illness or unstable medical condition;
* upper limb contusions, fractures (based on the imaging examination) or flaccid paralysis (by using noxious stimuli to upper limbs, motor sub-scale scores <1).

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
The level of consciousness in DOC patients | Within 2 days
  All patients were classified as the MCS and VS by the Coma recovery scale-revised

CONTACTS AND LOCATIONS:
Overall Officials: Haibo Di, Pro., Study Chair — International Vegetative State and Consciousness Science Institute, Hangzhou Normal University
Locations (1):
- International Vegetative State and Consciousness Science Institute, Hangzhou Normal University, Hangzhou, Zhejiang, China